CLINICAL TRIAL: NCT02896283
Title: The Effect of Low-Level Laser Therapy on Patient's Pain and Healing of Palatal Donor Site Following Free Gingival Graft: A Randomized Controlled Clinical Trial
Brief Title: Effect of Low-Level Laser on Pain and Healing of Donor Site Following Free Gingival Graft
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Neda Moslemi, Assistant Professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 91-01-97-16886
Record Dates: First submitted 2012-12-15; First posted 2016-09-12 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Gingival Recession
Keywords: wound healing; low-level laser therapy; gingival recession
MeSH Terms: conditions — Gingival Recession | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low-level laser therapy (Experimental): Low-level laser (Diode, 66o nanometer, power:200 milli Watt (mW), Continuous wave, time of irradiation:32 seconds)is irradiated in donor site
  Interventions: Radiation: Low-level laser therapy
- Turned-off laser (Placebo Comparator): The same protocol is applied in te donor site, unless the laser is remained off.
  Interventions: Radiation: Turned-off laser

INTERVENTIONS:
Radiation: Low-level laser therapy — Low-level laser therapy with the following parameters: Wavelength:660 nanometer, power: 200 mW, continuous mode, tme of irradiation: 32 seconds
  Other Names: low-level laser
  Arms: low-level laser therapy
Radiation: Turned-off laser — Laser device is turned-off. All parameters are like experimental group, however the laser in turned-off.
  Other Names: Placebo
  Arms: Turned-off laser

SUMMARY:
The aim of this randomized split-mouth design clinical trial is to clinically evaluate the effectiveness of diode laser in the healing of donor site of palate in free gingival graft.

DETAILED DESCRIPTION:
Free gingival graft is the most predictable and successful method for increasing the width of keratinized tissue around teeth/dental implants and vestibular deepening. However, patient discomfort during the healing time is a major disadvantage of this procedure. Several methods have been introduced to accelerate the healing time and reduction of patient's pain during first days after surgery. Low-level lasers have shown promising results in biostimulation of cell growth and differentiation in cultures. However, there are lack of well designed double blind placebo controlled randomized controlled clinical studies evaluating the effects of Low-level laser therapy in acceleration of wound healing and pain relief of patients undergoing free gingival grafts.

ELIGIBILITY:
Inclusion Criteria:

* lack of keratinized tissue around teeth (bilateral)

Exclusion Criteria:

* patients with systemic diseases
* non-cooperative patients
* smokers
* poor oral hygiene
* root surface restorations or active caries

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
degree of epithelialization | At day 7
  3% hydrogen peroxide (H2O2) was applied to the wound by a sterile gause to see the bubbling
  * Complete epithelialization: bubble was not seen
  * Partial epithelialization: bubbles were seen in lesser than half of donor site
  * No epithelialization: bubble were seen in more than half of donor site
degree of epithelialization | At day 14
  3% hydrogen peroxide (H2O2) was applied to the wound by a sterile gause to see the bubbling
  * Complete epithelialization: bubble was not seen
  * Partial epithelialization: bubbles were seen in lesser than half of donor site
  * No epithelialization: bubble were seen in more than half of donor site
degree of epithelialization | At day 21
  3% hydrogen peroxide (H2O2) was applied to the wound by a sterile gause to see the bubbling
  * Complete epithelialization: bubble was not seen
  * Partial epithelialization: bubbles were seen in lesser than half of donor site
  * No epithelialization: bubble were seen in more than half of donor site

SECONDARY OUTCOMES:
Visual analogue scale (VAS) pain score | at day 1
  ask from patient about numbers of tablet consumption,record VAS analysis
Visual analogue scale (VAS) pain score | at day 2
  ask from patient about numbers of tablet consumption,record VAS analysis
Visual analogue scale (VAS) pain score | at day 3
  ask from patient about numbers of tablet consumption,record VAS analysis
Visual analogue scale (VAS) pain score | at day 4
  ask from patient about numbers of tablet consumption,record VAS analysis
Visual analogue scale (VAS) pain score | at day 5
  ask from patient about numbers of tablet consumption,record VAS analysis
Visual analogue scale (VAS) pain score | at day 6
  ask from patient about numbers of tablet consumption,record VAS analysis
Visual analogue scale (VAS) pain score | at day 7
  ask from patient about numbers of tablet consumption,record VAS analysis
Visual analogue scale (VAS) pain score | at day 14
  ask from patient about numbers of tablet consumption,record VAS analysis
Clinical healing | at day 1
  Photographs were taken from donor and recipient sites. Three expert blinded periodontist photographs photographs based on shade,morphology and texture at two sessions by 48 hours interval.
Clinical healing | at day 2
  Photographs were taken from donor and recipient sites. Three expert blinded periodontist photographs photographs based on shade,morphology and texture at two sessions by 48 hours interval.
Clinical healing | at day 7
  Photographs were taken from donor and recipient sites. Three expert blinded periodontist photographs photographs based on shade,morphology and texture at two sessions by 48 hours interval.
Clinical healing | at day 14
  Photographs were taken from donor and recipient sites. Three expert blinded periodontist photographs photographs based on shade,morphology and texture at two sessions by 48 hours interval.
Clinical healing | at day 21
  Photographs were taken from donor and recipient sites. Three expert blinded periodontist photographs photographs based on shade,morphology and texture at two sessions by 48 hours interval.

CONTACTS AND LOCATIONS:
Overall Officials: Neda Moslemi, Study Director — Laser Research Center of Dentistry, Tehran University of Medical Sciences
Locations (1):
- Neda Moslemi, Tehran, Tehran Province, Iran